CLINICAL TRIAL: NCT03033797
Title: Augmentative and Alternative Communication in Games With Virtual Reality in Intellectual Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Regiani Guarnieri, Graphic Computer Specialist, Faculdade de Medicina do ABC
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 54172416.6.0000.0082
Record Dates: First submitted 2017-01-20; First posted 2017-01-27 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Intellectual Disability
Keywords: assitive technology; virtual reality games; intellectual disability; augmentative and alternative communication
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MoviLetrando-MoveHero (Experimental): Half of the children will play first two different levels of the game MoviLetrando (2 minutes each) and, after the game MoveHero, more 2 minutes
  Interventions: Device: MoviLetrando; Device: MoveHero
- MoveHero-MoviLetrando (Experimental): The other half of the children will play first 2 minutes of the game MoveHero and after, two different levels of the Game MoviLetrando, two minutes each.
  Interventions: Device: MoviLetrando; Device: MoveHero

INTERVENTIONS:
Device: MoviLetrando — Half of the participants will play two different levels of the Game MoviLetrando, two minutes each.
Device: MoveHero — Half of the participants will play 2 minutes of the game MoveHero.

SUMMARY:
Background: Games using motion capture from webcam have become increasingly popular. A population that lacks much stimulus in the teaching-learning process has under-explored the benefits of this kind of games: The Intellectually Disabled. The aim of this study is to analyse the effectiveness of games with virtual reality in the total reaction time. Method: A convenience sample of 165 Intellectually Disabled participants will have their performance measured using a virtual reality game. The intervention is to play two different games twice, in two sessions with an interval of, at least, seven days between the sessions. Participants will be randomized between two raters, both master students.

ELIGIBILITY:
Inclusion Criteria:

* All the children that uses to go the institution where the data collection will be realised (APAE).

Exclusion Criteria:

* Those who decline to participate
* Those who are not present in the two days of evaluation.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Estimated)
Dates: Start 2016-03-08 (Actual); Primary Completion 2018-03-10 (Estimated); Study Completion 2018-03-24 (Estimated)

PRIMARY OUTCOMES:
total reaction time | 6 minutes
  decrease in time indicates a better performance

SECONDARY OUTCOMES:
time MoviLetrando | up to 15 days
  less time to hit the targets indicates a better performance
acerts MoviLetrando | up to 15 days
  more hits indicates a better performance

CONTACTS AND LOCATIONS:
Locations (1):
- Associação de Pais e Amigos dos Excepcionais, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No